CLINICAL TRIAL: NCT00442247
Title: A Randomised, Controlled Study of Bimesh, Pelvicol for Vaginal Wall Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Feb-UH-2007
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Vaginal Prolapse
Keywords: anterior vaginal wall prolapse, Pelvicol, biomesh; Anterior vaginal wall prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pelvicol

SUMMARY:
Anterior vaginal wall prolapse is a common problem. Until now many different surgical techniques have been evaluated but so far recurrence is often still observed. Therefore, synthetic mesh or biomesh for vaginal prolapse reconstruction have been introduced.

DETAILED DESCRIPTION:
Anterior vaginal wall prolapse is a common problem. Until now many different surgical techniques have been evaluated but so far recurrence is often still observed. Therefore, synthetic mesh or biomesh for vaginal prolapse reconstruction have been introduced. However, is is now known whether these methods are superior to the replication of the pubocervicale fascia, a method which is well described and have been used for many years. Furthermore, most studies evaluating the used of mesh for anterior vaginal wall prolapse have not been controlled studies and been irrespective to whether the repair was a primary or secondary operation.

ELIGIBILITY:
Inclusion Criteria:

* Anterior vaginal wall prolapse greater than grade 2 ICS qualifications, International Continence Society Committee for Standardisation of Terminology

Exclusion Criteria:

* Recurrent vaginal prolapse, wault prolapse

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2008-12

PRIMARY OUTCOMES:
Difference in POP-Q measurements for vaginal prolapse

SECONDARY OUTCOMES:
Affect on bladder function after surgery for anterior vaginal wall prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Hviid, MD, Principal Investigator — Roskilde County Hospital, Dept. of Obstetrics and Gynecology, Roskilde University Hospital, Denmark
Locations (1):
- Dept. of Obstetrics and Gynecology, Roskilde, Denmark